CLINICAL TRIAL: NCT03809962
Title: Efficacy and Safety of Ostenil® Plus in the Treatment of Coxarthrosis
Status: Completed | Type: Observational
Sponsor: TRB Chemedica AG (Industry)
Responsible Party: Sponsor
Other Study IDs: OSTH-PMCF-DE-2018-01
Record Dates: First submitted 2019-01-14; First posted 2019-01-18 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Coxarthrosis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ostenil® Plus: 1-3 injections of sodium hyaluronate 2% (40 milligrams (mg) / 2,0 millilitres (ml)) in weekly interval.
  Interventions: Device: Ostenil® Plus

INTERVENTIONS:
Device: Ostenil® Plus — Ostenil® Plus is a CE-certified viscoelastic solution for injection into the Joint cavity, containing 2.0 % Sodium hyaluronate from fermentation

SUMMARY:
PMCF study to observe the Routine application of Ostenil® Plus in the Treatment of pain and restricted mobility in degenerative and traumatic changes of the Hip Joint.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 18 years of age and in good general health condition
2. Signed informed consent
3. Existing Ostenil® Plus recommendation for the treatment of coxarthrosis

Exclusion Criteria:

1. Known hypersensitivity to one of the OSTENIL® PLUS components
2. Known pregnancy or lactating females
3. Previous/concomitant participation in clinical investigation within the last 3 months prior to study inclusion
4. Subjects not capable of contracting and of understanding the nature, risks, significance and implications of the clinical investigation and unable to form a rational intention in the light of these facts
5. Subjects unable to understand informed consent or having a high probability of non compliance to the study procedures and / or non completion of the study according to investigator's judgement (e.g. illiteracy, insufficient knowledge of local language)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Coxarthrosis and a Recommendation for Treatment with Ostenil® Plus.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Change of Pain Intensity compared to Baseline (VAS-slider) | Day 7, Day 14, Day 84 after last injection, Day 168 after last injection
  Evaluation of Pain Intensity by the Patient on a 10 cm VAS-slider (10 cm equals the most pain)
Change of Range of Motion compared to Baseline (Goniometer measurement) | Day 7, Day 14, Day 84 after last injection, Day 168 after last injection
  Assessment of the Range of internal and exernal rotation of the Hip Joint using a Goniometer.
Change of Subjective Symptom Evaluation (Overall Impression on a scale from 1 to 5) | Day 7, Day 14, Day 84 after last injection, Day 168 after last injection
  The Change of Overall Subjective Symptom Evaluation on a scale from 1 (much improved) to 5 (much worse).
Incidence of Treatment-Emergent Adverse Events | Up to Day 252 after the last injection
Change of Subjective Therapy Evaluation of Pain (HOOS Questionnaire) compared to Baseline | Day 84 after last injection, Day 168 after last injection
  Hip Disability and Osteoarthritis Outcome Score (HOOS) to assess Pain on a 5-point Likert scale
Change of Subjective Therapy Evaluation of Stiffness (HOOS Questionnaire) compared to Baseline | Day 84 after last injection, Day 168 after last injection
  Hip Disability and Osteoarthritis Outcome Score (HOOS) to assess Stiffness on a 5-point Likert scale
Change of Subjective Therapy Evaluation of Function in daily living (HOOS Questionnaire) compared to Baseline | Day 84 after last injection, Day 168 after last injection
  Hip Disability and Osteoarthritis Outcome Score (HOOS) to assess Function in daily living on a 5-point Likert scale
Change of Subjective Therapy Evaluation of Quality of Life (HOOS Questionnaire) compared to Baseline | Day 84 after last injection, Day 168 after last injection
  Hip Disability and Osteoarthritis Outcome Score (HOOS) to assess Quality of Life on a 5-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Knut Behle, Dr. med., Principal Investigator — OrthopädieZentrum Maschen; Darja Becker, Dr. med., Principal Investigator — Orthopädie Praxis Dr. Darja Becker
Locations (7):
- Germany (7):
  - Orthopädische Praxis Rahlstedt, Hamburg, Hamburg
  - Gemeinschaftspraxis für Orthopädie und Unfallchirurgie, Bad Oldesloe, Schleswig-Holstein
  - Orthopraxis Kiel, Gettorf, Schleswig-Holstein
  - Zentrum für Medizin des Bewegungsapparates, Heide, Schleswig-Holstein
  - Orthopädische Gemeinschaftspraxis Eutin, Eutin
  - Orthopädie Praxis, Ramelsloh
  - OrthopädieZentrum Maschen, Seevetal